CLINICAL TRIAL: NCT05787691
Title: Enhanced vs. Standard Pain Management of Patients at Risk for Chronic Post-surgical Pain: a Randomized Controlled Pilot Trial
Brief Title: Enhanced vs.Standard Pain Management of Patients at Risk for Chronic Post-surgical Pain
Acronym: ALDOpilot
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Paulina Sypniewska El Khoury, MD, Principal Investigator, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UGeneva 20221005
Record Dates: First submitted 2023-02-07; First posted 2023-03-28 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Chronic Post Surgical Pain
Keywords: total knee prothesis; spine surgery; thorax surgery; transitional pain service
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individualised Pain Management (Experimental): In the intervention group, patients will be followed by the team of the "transitional pain service" of the HUG, and depending on individual risk factors, contraindications and following discussion with the patient (shared decision-making) the bundle of individually targeted measures will be applied.
  Interventions: Other: Individualised pain management
- Standard care (No Intervention): In the control group, no specific measures will be applied, and patients are followed by their surgeon and general practitioner. In addition, during the hospitalization the Acute Pain Team may be requested. In case of persistent pain, it may happen that the surgeon or the general practitioner refers a patient to a chronic pain specialist.

INTERVENTIONS:
Other: Individualised pain management — TPS pain management consists in an evaluation by a pain physician, followed by specific measures for patients identified as having a particularly high risk of CPSP. The choice of these measures will be individualised according to specific risk factors and left to the discretion of the pain physician.
  Potential measures: patient education, adjustment of analgesic therapy, referral to a psychiatrist or psychologist, cognitive behavioural therapy, hypnosis, use of locoregional analgesia for surgery, infusions of ketamine and/or lidocaine, introduction of gabapentins and/or antidepressants.
  Other Names: Transitional Pain Service TPS
  Arms: Individualised Pain Management

SUMMARY:
The goal of this pragmatic pilot clinical trial is to test the feasibility of the trial in terms of the number of patients recruited in a given period.

The main question it aims to answer is to assess the number of eligible patients and number of patients willing to participate per month.

Participants will be followed either by the team of "transitional pain service" (intervention group) or by a surgeon or the general practitioner (standard care). Depending on individual risk factors, patients in the intervention group will be offered some targeted measures, for example:

* hypnosis,
* patient education,
* evaluation by psychiatrist,
* psychotherapy,
* locoregional anesthesia,
* anti-depressant treatment Participants (in both intervention and standard care groups) will be asked to answer some questions before surgery, during the first week following the surgery and six months after the surgery.

DETAILED DESCRIPTION:
Moderate to severe persistent post-surgery pain occurs in up to 12% of patients at 6 months post-surgery according to the large European study cohort. Our own data from a previous study at the University Hospitals of Geneva (HUG) (unpublished, alerte douleur-ALDO study) showed a prevalence of chronic post-surgical pain (CPSP) 6 months after selected types of surgery of 30.9%. Strategies to detect and prevent CPSP have not been applied systematically in clinical practice until now, despite routine surgical follow-up visits after surgery.

There are only few hospitals who have implemented a "transitional pain service (TPS)" to diminish the risk of the transition of acute to chronic pain after surgery, and the Anesthesia Department of the University Hospitals of Geneva is currently experimenting with such a team. A future study needs to validate the effectiveness of this approach.

The present study is planned as a pilot trial to test the feasibility, usability, acceptance, and to provide the parameters necessary to design this future study validating or refuting the utility of individually targeted combinations of preventive measures implemented by a "transitional pain service" in reducing the incidence of chronic pain 6 months after surgery.

The primary objective is to evaluate the feasibility of the trial in terms of the number of patients recruited in a given period.

Secondary objectives are:

* To determine patient acceptance of the proposed interventions and thus the percentage of patients receiving the planned interventions in reality in the treatment group
* To determine the percentage of patients in the control group receiving the treatments proposed in the intervention group by other caregivers outside of the study (patients in the control group may even receive such treatment by the investigators if requested by the patients or another physician)
* To evaluate the usefulness of a transitional pain service (TPS) from a patient perspective
* To determine the optimal primary outcome measure of the definitive trial

The study is a single-center, randomized controlled clinical pilot trial, designed to estimate the parameters necessary for planning a definitive, potentially multicentric study.

The randomization will follow 1: 1 allocation, with 2 parallel groups of patients with increased risk for CPSP (intervention group vs. a group with a routine follow up). A total of 60 patients will be included.

Patients undergoing spinal surgery, total knee replacement surgery or thoracic surgery will be screened for inclusion in the study.

Patients will be contacted for an informed consent, either by telephone and email, or by a personal visit before the surgery.

Following informed consent, all patients included will receive a set of questionnaires (by email or in paper form) concerning psychological risk factors and details about preexisting chronic pain.

Consenting patients will be randomized using a computer-generated list to either the treatment or the control group.

In neither group, surgical management of included patients will be influenced by the study.

In the intervention group, patients will be followed by the team of the "transitional pain service" of the University Hospitals of Geneva, and depending on individual risk factors, contraindications and following discussion with the patient (shared decision-making) the bundle of individually targeted measures.

In the control group, no specific measures will be applied, and patients are followed by their surgeon and general practitioner. In addition, during the hospitalization the Acute Pain Team may be requested. In case of persistent pain, it may happen that the surgeon or the general practitioner refers a patient to a chronic pain specialist. This will not lead to the exclusion of the patient.

Patients of both groups will receive identical follow-up questionnaires after surgery and outcome questionnaires by electronic or written form at 6 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for spine surgery or total knee replacement surgery or thoracic surgery
* patients of 18 years or more
* ability to speak and read French

Exclusion Criteria:

* inability to consent and to follow the procedures of the study
* emergency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05-12 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
recruitment rate | 6 months
  number of patients included in the study per month

SECONDARY OUTCOMES:
Retention rate | 6 months
  number of patients who complete the study
Data completeness rate | 6 months
  number of patients with complete data sets
Number of measures accepted at 6 months | 6 months
  Number of patients who accepted each preventive measure in the intervention and control groups
Number of measures completed at 6 months | 6 months
  Number of patients who completed each preventive measure in the intervention and control groups
Usefulness of a "transitional pain service" (TPS) from a patient perspective | 6 months
  number of patients evaluating the preventive treatment useful or non-useful at 6 months post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Paulina Sypniewska El Khoury, MD, Principal Investigator — University Hospital, Geneva
Locations (1):
- Hôpitaux Universitaires de Genève, Geneva, Switzerland